CLINICAL TRIAL: NCT06621940
Title: Effect of High Protein Diet on Total Antioxidant Capacity
Brief Title: Effect of Proteins on Antioxidant Capacity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Aslı Onur Canaydın, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ERU-BES-AOC-02
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: High Protein Dietary Intake
Keywords: High protein diet; Antioxidant capacity; Oxidative stress; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: It consists of two parallel groups receiving a high-protein diet and a normal-protein diet.
Who Masked: Participant
Masking Description: The content of the diet will be given to the participants without specifying it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein Diet (Experimental): The energy composition of the high protein diet will be calculated as 40% carbohydrate, 30% protein and 30% fat. It will be stated that individuals should not eat anything other than the foods to be sent during the weeks of the diet.
  Interventions: Other: High Protein Diet
- Normal Protein Diet (Experimental): The energy composition of the high protein diet will be calculated as 55% carbohydrate, 15% protein and 30% fat. It will be stated that individuals should not eat anything other than the foods to be sent during the weeks of the diet.
  Interventions: Other: Normal Protein Diet

INTERVENTIONS:
Other: High Protein Diet — Individuals will be placed on a high protein diet for 10 days.
  Arms: High Protein Diet
Other: Normal Protein Diet — Individuals will be placed on a normal protein diet for 10 days.
  Arms: Normal Protein Diet

SUMMARY:
This study was planned to provide information about the effect of short-term high protein diet (HPD) feeding on early antioxidant response in women. The definition of HPDs cannot be determined exactly. It is defined differently by various scientific authorities. However, protein is targeted to be approximately 30% of total energy in HPD. It has been determined that HPDs increase satiety, thermogenesis, and provide body weight loss and maintenance of loss. In general, there is evidence that HPD provides more body weight loss in a short time compared to low protein diets. It has been emphasized that the effect of high protein diet on weight loss is related to creating satiety, thus decreasing food intake and increasing thermogenesis. However, the physiological, biochemical and molecular events that occur due to HPD feeding have not been fully understood and the results have not been explained. The effects of HPDs have been determined to last from 1 to 6 days to 6 months. The absence of any study in the literature on the short-term and long-term effects of HPD on oxidative events in humans reveals the original value of this study. Therefore, considering that long-term HPD feeding may increase the risk of cardiovascular disease, blood pressure, and blood lipid levels, the effect of short-term HPD feeding on antioxidant capacity will be investigated in order to avoid these side effects. The planned interviews and measurements for this prospective analytical study will be carried out in the Anthropometry laboratory of the Department of Nutrition and Dietetics, Faculty of Health Sciences at Erciyes University, and blood analyses will be carried out in the Betül Ziya Eren Genome and Stem Cell Research Center laboratory and the Erciyes University Gülser and Dr. Mustafa Gündoğdu Comprehensive Service Laboratory. Healthy female individuals will be applied HPD for 10 days and a normal diet for 10 days as a control. As a result of the applied diets, the expected results of the study are that HPD will cause a decrease in body weight and an increase in lean body mass, even for a short time, and that HPD will have an effect on diet-induced inflammation, cause oxidative stress, affect antioxidant capacity and cause changes in the measured parameters.

DETAILED DESCRIPTION:
Today, most individuals try various nutritional models/diets to reduce body weight. One of the most popular of these diets is the diets that reduce carbohydrate intake. Western societies generally avoid high carbohydrates and fat intake. For this reason, interest in high protein intake in diets is increasing day by day. Although there is no general consensus on what a high-protein diet is, the high protein diet (HPD) applied for weight loss studies is diets that contain approximately 30% of the energy provided by protein. The World Health Organization (WHO) has defined obesity as an endemic public problem and stated that its prevalence is increasing. With the increase in obesity, individuals try various dietary modifications to achieve weight loss. These include diets with a more regular macro and micronutrient pattern, such as the Mediterranean Diet and the DASH diet, and diets that may cause deficiencies in terms of macro and micronutrients, such as Atkins, South Beach, Zone, and Stillman, which contain high protein. The most important reasons why high-protein diets attract attention are that they cause rapid weight loss and provide satiety. This positive effect of HPDs on weight loss has attracted the attention of dietitians and caused them to increase the protein ratio in diets. Scientific authorities against popular diets; what is really known about popular diets, the scientific nature of the information, whether it is effective in maintaining body weight, if it is effective, its effect on body composition, micronutrient level, metabolic indicators, hunger-satiety, psychological state, chronic disease risk, its effect on leptin and insulin levels, which provide hormone regulation in long-term energy intake and expenditure.

It is known that HPDs provide more effective results in body weight loss compared to low protein diets. It is suggested that this effect occurs as a result of increased thermogenesis, increased satiety and suppressed appetite, and reduced glycemic index and glycemic load due to the replacement of refined carbohydrates with proteins. In addition to this positive effect on weight loss, there are possible short- and long-term side effects of HPD nutrition. Known complications of long-term HPD nutrition include increased cardiovascular disease risk, blood pressure, blood lipids, and kidney dysfunction. Cardiovascular problems in particular are a source of concern because they will counteract the short-term positive effect of HPD on weight loss and increase the burden of cardiovascular disease in the long term. Studies generally focus on HPD and weight loss; there is limited data on the relationship between HPD nutrition and metabolic dysfunction such as endothelial dysfunction, inflammatory markers, antioxidant status, and other chronic diseases. The physiological, biochemical, and molecular events that occur due to high protein diet nutrition have not been fully understood and their results have not been explained.

High protein diets (especially low carbohydrate diets) are thought to have negative effects because they cause a decrease in fruit and vegetable consumption. In those who eat a HPD, especially inadequate vitamin A, C and E in their diets, this will have a negative effect on antioxidant systems and will pave the way for the development of many chronic and metabolic diseases in the long term. Despite the positive effects of HPD applied as a weight loss diet in the short term, it is thought that the oxidative stress and inflammation it will create in the long term will cause an increase in chronic and metabolic diseases as well as comorbidities. This increase in the disease burden will increase health expenditures both individually and socially.

Therefore, this study was planned to provide information about the effect of short-term HPD feeding on early antioxidant response in adult, healthy, normal body mass index female individuals. As a result of the study, it is thought that short-term HPD feeding will cause an increase in oxidative stress, a decrease in antioxidant capacity and an increase in inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Being between 19-45 years of age,
* Not changing physical activity throughout the study,
* Having a BMI of 18.5-24.9 kg/m2,
* Being healthy

Exclusion Criteria:

* Having a BMI of <18.5 and ≥25 kg/m2,
* Having a chronic disease,
* Smoking and drinking alcohol,
* Using vitamin-mineral supplements and herbal supplements,
* Being pregnant or breastfeeding,
* Having entered menopause,
* Being on any diet.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Antioxidant capacity after high protein diet | Day after diet end
  After the diet, antioxidant biomarkers [antioxidant status (TAS), total oxidant status (TOS)] will be measured in the blood. Lower values represent a worse outcome.
Anthropometric measurements after high protein diet | Day after diet end
  Anthropometric measurements will be made after the diet. An increase in anthropometric measurements represents a worse result.

IPD SHARING:
Plan to Share IPD: No